CLINICAL TRIAL: NCT02395133
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Investigating the Efficacy and Safety of Multiple Dupilumab Dose Regimens Administered as Monotherapy for Maintaining Treatment Response in Patients With Atopic Dermatitis
Brief Title: A Study to Confirm the Efficacy and Safety of Different Dupilumab Dose Regimens in Adults With Atopic Dermatitis (AD)
Acronym: SOLO-CONTINUE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R668-AD-1415; 2014-003384-38 (EudraCT Number)
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-02

CONDITIONS: Atopic Dermatitis
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Subcutaneous injection of Placebo (for Dupilumab) was administered once weekly (QW) from Week 1 (Day 1) to Week 36.
  Interventions: Drug: Placebo
- Dupilumab 300 mg Q8W (Experimental): Subcutaneous injection of Dupilumab 300 milligram (mg) alternatively with placebo (matched to Dupilumab) was administered once every eight week (Q8W) from Week 1 to Week 36.
  Interventions: Drug: Dupilumab
- Dupilumab 300 mg Q4W (Experimental): Subcutaneous injection of Dupilumab 300 mg alternatively with placebo (matched to Dupilumab) was administered once every four week (Q4W) from Week 1 to Week 36.
  Interventions: Drug: Dupilumab
- Dupilumab 300 mg Q2W/QW (Experimental): Subcutaneous injection of Dupilumab 300 mg alternatively with placebo (matched to Dupilumab) was administered once every week (QW) or twice a week (Q2W) from Week 1 to Week 36.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Subcutaneous injection of Dupilumab 300 mg alternatively with placebo (matched to Dupilumab) was administered.
  Other Names: REGN668; SAR231893
  Arms: Dupilumab 300 mg Q2W/QW; Dupilumab 300 mg Q4W; Dupilumab 300 mg Q8W
Drug: Placebo — Subcutaneous injection of Placebo (for Dupilumab) was administered once weekly (QW).
  Arms: Placebo

SUMMARY:
The primary objective of the study was to assess the ability of different Dupilumab dose regimens, administered as monotherapy, to maintain the treatment response achieved after 16 weeks of initial treatment with Dupilumab monotherapy compared to placebo.

ELIGIBILITY:
Key Inclusion Criteria:

1. Must have completed the treatment phase in 1 of the two 16-week initial treatment studies (R668-AD-1334 or R668-AD-1416).
2. Must have achieved at least 1 of the following 2 treatment success criteria:

   Investigator Global Assessment (IGA) = 0 or 1 (clear or almost clear) at week 16 OR Eczema Area and Severity Index >= 75% (EASI-75) (at least 75% reduction in EASI score from baseline to week 16)
3. Must be willing and able to comply with clinic visits and study-related procedures
4. Must provide signed informed consent
5. Must be able to understand and complete study-related questionnaires

Key Exclusion Criteria:

1. Receipt of rescue medication for AD in the initial treatment study
2. Any conditions that require permanent discontinuation of study treatment in either initial treatment study
3. Planned or anticipated major surgical procedure during the participants's participation in this study
4. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during this study
5. Women unwilling to use adequate birth control, if of reproductive potential* and sexually active. Adequate birth control is defined as agreement to consistently practice an effective and accepted method of contraception, whenever engaging in heterosexual intercourse, throughout the duration of the study and for 120 days after last dose of study drug. These include hormonal contraceptives, intrauterine device, or double barrier contraception (e.g, condom + diaphragm), or a male partner with documented vasectomy. Additional requirements for acceptable contraception may apply in certain countries, based on local regulations. Investigators in these countries will be notified accordingly in a protocol clarification letter.

(*For females, menopause is defined as at least 12 consecutive months without menses; if in question, a follicle stimulating hormone level of >= 25 milli units per milliliter (mU/mL) must be documented. Hysterectomy, bilateral oophorectomy, or bilateral tubal ligation must be documented, as applicable; if documented, women with these conditions are not required to use additional contraception).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals

REFERENCES:
- [Derived] Stander S, Yosipovitch G, Simpson EL, Kim BS, Kabashima K, Thaci D, Metz M, Chen Z, Hagen S, Bastian M. Onset and Long-Term Maintenance of Optimal Itch Response in Adult Patients with Moderate-to-Severe Atopic Dermatitis Treated with Dupilumab: Post Hoc Analysis from Two Phase 3 Trials. Adv Ther. 2025 Apr;42(4):1800-1810. doi: 10.1007/s12325-025-03124-8. Epub 2025 Feb 19. PMID 39969783
- [Derived] Kamal MA, Kosloski MP, Lai CH, Partridge MA, Rajadhyaksha M, Kanamaluru V, Bansal A, Shabbir A, Shumel B, Ardeleanu M, Richards SM, Yan H, Xu CR, Rodriguez-Marco A, Xiao J, Khokhar FA, Gherardi G, Babilonia E, Maloney J, Mortensen E, Akinlade B, Braunstein N, Stahl N, Torri A, Davis JD, DiCioccio AT. Immunogenicity of dupilumab in adult and pediatric patients with atopic dermatitis. Front Immunol. 2024 Nov 11;15:1466372. doi: 10.3389/fimmu.2024.1466372. eCollection 2024. PMID 39588375
- [Derived] Worm M, Simpson EL, Thaci D, Bissonnette R, Lacour JP, Beissert S, Kawashima M, Ferrandiz C, Smith CH, Beck LA, Chan KC, Chen Z, Akinlade B, Hultsch T, Staudinger H, Gadkari A, Eckert L, Davis JD, Rajadhyaksha M, Graham NMH, Pirozzi G, Stahl N, Yancopoulos GD, Ardeleanu M. Efficacy and Safety of Multiple Dupilumab Dose Regimens After Initial Successful Treatment in Patients With Atopic Dermatitis: A Randomized Clinical Trial. JAMA Dermatol. 2020 Feb 1;156(2):131-143. doi: 10.1001/jamadermatol.2019.3617. PMID 31876900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 15 countries between 25 March 2015 and 18 October 2016. A total of 422 participants were randomized in the study.
Pre-assignment Details: Out of the 475 participants, 422 were randomized and 420 received either placebo or Dupilumab. Participants were randomized in 2:1:1:1 ratio to receive Dupilumab 300 milligram (mg) once weekly/twice weekly (QW/Q2W), Dupilumab 300 mg four times a week (Q4W), Dupilumab 300 mg eight times a week (Q8W) and Placebo.
Groups:
- Placebo QW: Subcutaneous injection of Placebo (for Dupilumab) was administered weekly (QW) from Week 1 (Day 1) to Week 36.
- Dupilumab 300 mg Q8W: Subcutaneous injection of Dupilumab 300 mg alternatively with placebo (matched to Dupilumab) once every eight week (Q8W) from Week 1 to Week 36.
- Dupilumab 300 mg Q4W: Subcutaneous injection of Dupilumab 300 mg alternatively with placebo (matched to Dupilumab) once every four week (Q4W) from Week 1 to Week 36.
- Dupilumab 300 mg Q2W/QW: Subcutaneous injection of Dupilumab 300 mg alternatively with placebo (matched to Dupilumab) once every week (QW) or twice a week (Q2W) from Week 1 to Week 36.
Period: Overall Study
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Started (Full Analysis Set (FAS) included all randomized participants) | 83 | 84 | 86 | 169
Completed | 69 | 75 | 76 | 155
Not Completed | 14 | 9 | 10 | 14
Not completed — Adverse Event | 4 | 1 | 3 | 0
Not completed — Lack of Efficacy | 1 | 0 | 1 | 1
Not completed — Protocol Violation | 1 | 1 | 0 | 3
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Pregnancy | 0 | 0 | 3 | 0
Not completed — Consent withdrawn with no reason given | 1 | 3 | 0 | 2
Not completed — Consent withdrawn with personal reason | 0 | 1 | 0 | 3
Not completed — Sponsor decision | 2 | 0 | 0 | 1
Not completed — Other than specified above | 5 | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW | Total
Number analyzed (Participants) | 83 | 84 | 86 | 169 | 422
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.1 (13.64) | 37.3 (13.98) | 38.5 (16.76) | 38.5 (13.94) | 38.2 (14.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 43 | 87 | 195
  Male | 51 | 51 | 43 | 82 | 227
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 10 | 16
  Not Hispanic or Latino | 75 | 81 | 85 | 155 | 396
  Unknown or Not Reported | 6 | 0 | 0 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 17 | 18 | 16 | 31 | 82
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 8 | 4 | 7 | 26
  White | 54 | 56 | 64 | 124 | 298
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 2 | 7 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 38 | 39 | 38 | 77 | 192
  Japan | 12 | 11 | 12 | 23 | 58
  Europe | 33 | 34 | 36 | 69 | 172
Eczema Area and Severity Index (EASI) Score [Mean (Standard Deviation); unit: units on a scale] — The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points,with the higher scores reflecting the worse severity of AD.
  units on a scale | 2.5 (2.31) | 2.3 (2.33) | 2.8 (3.31) | 2.6 (2.92) | 2.6 (2.78)
Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) [Mean (Standard Deviation); unit: units on a scale] — Pruritus NRS scale is an assessment tool that is used to report the intensity of participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0= no itch; 10= worst itch imaginable]).
  units on a scale | 2.8 (2.11) | 2.7 (2.27) | 3.1 (2.16) | 2.8 (1.92) | 2.8 (2.08)
Body Surface Area (BSA) Involvement with AD [Mean (Standard Deviation); unit: percentage of body surface area] — Body surface area affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined.
  percentage of body surface area | 8.1 (8.21) | 7.9 (9.04) | 9.3 (10.51) | 7.9 (9.02) | 8.2 (9.18)
SCORing Atopic Dermatitis (SCORAD) Score [Mean (Standard Deviation); unit: units on a scale] — SCORAD was a clinical tool for assessing the severity of AD developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) were assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease).
  units on a scale | 16.8 (10.03) | 17.1 (9.41) | 17.5 (10.59) | 17.1 (10.49) | 17.1 (10.18)
Patient Oriented Eczema Measure (POEM) [Mean (Standard Deviation); unit: units on a scale] — The POEM was a 7-item questionnaire that assessed disease symptoms (dryness,itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]).
  units on a scale | 6.1 (5.43) | 6.8 (5.88) | 6.1 (5.11) | 6.4 (5.30) | 6.3 (5.40)
Dermatology Life Quality Index (DLQI) Score [Mean (Standard Deviation); unit: units on a scale] — The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL). The 10 questions assessed QOL over the past week, with an overall scoring of 0 (absent disease) to 30 (severe disease); a high score indicative of a poor QOL.
  units on a scale | 3.4 (4.25) | 3.0 (3.76) | 3.2 (3.93) | 3.4 (4.21) | 3.3 (4.06)
Total Hospital Anxiety Depression Scale (HADS) [Mean (Standard Deviation); unit: units on a scale] — The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression. Cut-offs for identifying psychiatric distress has been reported as 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression.
  units on a scale | 5.9 (6.36) | 7.1 (6.87) | 7.3 (7.53) | 6.4 (5.94) | 6.6 (6.53)

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Current Study Baseline and Week 36 in Percent Change in EASI From Parent Study Baseline (NCT02277743 and NCT02277769)
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Difference of percent change in EASI between current study baseline and week 36 in from parent study baseline (NCT02277743 and NCT02277769) was reported. Values after first rescue treatment used were set to missing before multiple imputation (MI).
Time Frame: Baseline (Parent Study), Baseline (Current Study) and Week 36 (Current study)
Population: The full analysis set (FAS) includes all randomized participants.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 83 | 84 | 86 | 169
percent change | 21.67 (3.134) | 6.84 (2.434) | 3.84 (2.283) | 0.06 (1.736)
Statistical Analysis 1: Comparison: Placebo QW vs Dupilumab 300 mg Q8W; A 2-sided hierarchical testing procedure was used for the co-primary and key secondary efficacy endpoints in a pre-specified order. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only when the previous endpoint was statistically significant at 0.05 level. Analysis was performed using ANCOVA method; Test type: Superiority; p = 0.0001, ANCOVA; Threshold for significance at 0.05 level; Percent Change Difference = -14.83, 95% CI 2-sided [-22.34 to -7.33]
Statistical Analysis 2: Comparison: Placebo QW vs Dupilumab 300 mg Q4W; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; Threshold for significance at 0.05 level; Percent Change Difference = -17.83, 95% CI 2-sided [-25.33 to -10.34]
Statistical Analysis 3: Comparison: Placebo QW vs Dupilumab 300 mg Q2W/QW; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; Threshold for significance at 0.05 level; Percent Change Difference = -21.61, 95% CI 2-sided [-28.36 to -14.87]

2. Primary Outcome: Percentage of Participants With Eczema Area and Severity Index >= 75% [EASI-75] at Baseline of Current Study Maintaining EASI-75 at Week 36
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-75 responders were the participants who achieved >=75% overall improvement in EASI score at Week 36. Values after first rescue treatment used were set to missing. Patients with missing value at week 36 were considered as a non-responder.
Time Frame: Week 36
Population: FAS population was used. Here, number of participants analyzed = participants with EASI-75 at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 79 | 82 | 84 | 162
percentage of participants | 30.4 | 54.9 | 58.3 | 71.6
Statistical Analysis 1: Comparison: Placebo QW vs Dupilumab 300 mg Q8W; Testing according to the hierarchical testing procedure (only performed if the previous endpoint was statistically significant). Analysis was performed using Cochran-Mantel-Haenszel test stratified by region, baseline disease severity and Dupilumab regimen received in parent studies; Test type: Superiority; p = 0.0040, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 24.5, 95% CI 2-sided [9.70 to 39.29]
Statistical Analysis 2: Comparison: Placebo QW vs Dupilumab 300 mg Q4W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 28.0, 95% CI 2-sided [13.32 to 42.58]
Statistical Analysis 3: Comparison: Placebo QW vs Dupilumab 300 mg Q2W/QW; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 41.2, 95% CI 2-sided [28.93 to 53.52]

3. Secondary Outcome: Percentage of Participants Maintaining Investigator Global Assessment (IGA) Response Within 1 Point of Baseline at Week 36
Description: IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear). Participants with IGA score of 0 or 1 at baseline and maintaining within 1 point of baseline were reported as responders. Values after first rescue treatment used were set to missing. Participants with missing value at a visit were considered as a non-responder.
Time Frame: Baseline, Week 36
Population: FAS population was used. Here, number of participants analyzed = participants with IGA 0 or 1 at Baseline from Interactive voice response system (IVRS).
Measure: Number; unit: percentage of participants
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 63 | 64 | 66 | 126
percentage of participants | 28.6 | 50.0 | 62.1 | 70.6
Statistical Analysis 1: Comparison: Placebo QW vs Dupilumab 300 mg Q8W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0130, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 21.4, 95% CI 2-sided [4.86 to 38.00]
Statistical Analysis 2: Comparison: Placebo QW vs Dupilumab 300 mg Q4W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 33.5, 95% CI 2-sided [17.38 to 49.72]
Statistical Analysis 3: Comparison: Placebo QW vs Dupilumab 300 mg Q2W/QW; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 42.1, 95% CI 2-sided [28.36 to 55.76]

4. Secondary Outcome: Percentage of Participants Maintaining Investigator Global Assessment (IGA) Response at 0 or 1 Point at Week 36
Description: IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear). Participants with IGA score of 0 or 1 at week 36 were reported as responders. Values after first rescue treatment were set to missing and participants with missing IGA scores at Week 36 were considered as non-responders.
Time Frame: Week 36
Population: FAS population was used. Here, number of participants analyzed = participants with IGA 0 or 1 at Baseline from IVRS.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 63 | 64 | 66 | 126
percentage of participants | 14.3 | 32.8 | 43.9 | 54.0
Statistical Analysis 1: Comparison: Placebo QW vs Dupilumab 300 mg Q8W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0209, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 18.5, 95% CI 2-sided [4.14 to 32.91]
Statistical Analysis 2: Comparison: Placebo QW vs Dupilumab 300 mg Q4W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0007, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 29.7, 95% CI 2-sided [14.89 to 44.42]
Statistical Analysis 3: Comparison: Placebo QW vs Dupilumab 300 mg Q2W/QW; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = 39.7, 95% CI 2-sided [27.42 to 51.95]

5. Secondary Outcome: Percentage of Participants With Weekly Average of Peak Daily Pruritus Numerical Rating Scale (NRS) Score Increased by 3 or More Points From Baseline to Week 35
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Values after first rescue treatment were set to missing and participants with missing peak NRS at Week 35 were considered as non-responders.
Time Frame: Baseline up to Week 35
Population: FAS population was used. Here, number of participants analyzed = participants with NRS <= 7 at Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 80 | 81 | 83 | 168
percentage of participants | 70.0 | 55.6 | 49.4 | 33.9
Statistical Analysis 1: Comparison: Placebo QW vs Dupilumab 300 mg Q8W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1048, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = -14.4, 95% CI 2-sided [-29.21 to 0.32]
Statistical Analysis 2: Comparison: Placebo QW vs Dupilumab 300 mg Q4W; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0107, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = -20.6, 95% CI 2-sided [-35.32 to -5.89]
Statistical Analysis 3: Comparison: Placebo QW vs Dupilumab 300 mg Q2W/QW; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Percentage difference = -36.1, 95% CI 2-sided [-48.40 to -23.74]

6. Secondary Outcome: Time to First Event of Investigator's Global Assessment (IGA) >= 2 for Participants With IGA 0 or 1 at Baseline
Description: IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear).
Time Frame: Baseline up to Week 36
Population: FAS population was used. Here, number of participants analyzed = participants with IGA 0 or 1 at Baseline from IVRS.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 63 | 64 | 66 | 126
Days | 57 [56 to 58] | 85 [59 to 113] | 80 [55 to 85] | 114 [85 to 169]

7. Secondary Outcome: Percentage of Participants With Increased Investigator's Global Assessment (IGA) Score 3 or 4 at Week 36
Description: IGA is an assessment scale used to determine severity of AD and clinical response to treatment on a 5-point scale (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe) based on erythema and papulation/infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear). Values after first rescue treatment were set to missing and participants with missing IGA scores at Week 36 were considered as responders (i.e. having a increase 3 or 4 of IGA value).
Time Frame: Week 36
Population: FAS population was used. Here, number of participants analyzed = participants with IGA 0 or 1 at Baseline from IVRS.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 63 | 64 | 66 | 126
percentage of participants | 66.7 | 48.4 | 34.8 | 26.2

8. Secondary Outcome: Percentage of Participants With Eczema Area and Severity Index-50 (EASI-50) (>= 50% Reduction in EASI Score) at Week 36
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. EASI-50 responders were the participants who achieved >= 50% overall improvement in EASI score from baseline to Week 36. Values after first rescue treatment were set to missing and participants with missing EASI-50 scores at Week 36 were considered as non-responders.
Time Frame: Week 36
Population: FAS population was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 83 | 84 | 86 | 169
percentage of participants | 39.8 | 54.8 | 60.5 | 73.4

9. Secondary Outcome: Absolute Change From Baseline in Eczema Area and Severity Index (EASI) at Week 36
Description: The EASI score was used to measure the severity and extent of AD and measured erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score ranges from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD. Values after first rescue treatment were set to missing and participants with missing Values at Week 36 were imputed by using multiple imputation method.
Time Frame: Baseline, Week 36
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 83 | 84 | 86 | 169
units on a scale | 6.61 (0.799) | 1.75 (0.738) | 1.37 (0.735) | 0.09 (0.511)

10. Secondary Outcome: Absolute Change From Baseline in SCORing Atopic Dermatitis (SCORAD) Score at Week 36
Description: SCORAD is a clinical tool for assessing the severity of AD developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease). Values after first rescue treatment used were set to missing (censoring) before MI.
Time Frame: Baseline, Week 36
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 83 | 84 | 86 | 169
units on a scale | 18.61 (2.107) | 6.62 (2.010) | 2.25 (1.899) | 0.99 (1.350)

11. Secondary Outcome: Absolute Change From Baseline in Peak Daily Pruritus Numerical Rating Scale (NRS) Score at Week 35
Description: Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), both maximum and average intensity, during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]). Values after first rescue treatment used were set to missing before MI.
Time Frame: Baseline, Week 35
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 83 | 84 | 86 | 169
units on a scale | 2.5 (0.29) | 1.1 (0.27) | 0.6 (0.25) | -0.1 (0.20)

12. Secondary Outcome: Absolute Change From Baseline in Body Surface Area (BSA) Through Week 36
Description: BSA affected by AD was assessed for each section of the body (the possible highest score for each region was: head and neck [9%], anterior trunk [18%], back [18%], upper limbs [18%], lower limbs [36%], and genitals [1%]). It was reported as a percentage of all major body sections combined. Values after first rescue treatment used were set to missing (censoring) before MI.
Time Frame: Baseline through Week 36
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: meter square
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 83 | 84 | 86 | 169
meter square | 9.16 (1.642) | 2.74 (1.530) | 1.74 (1.457) | -1.27 (1.044)

13. Secondary Outcome: Absolute Change From Baseline Through in Patient Oriented Eczema Measure (POEM) Through Week 36
Description: The POEM is a 7-item questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) with a scoring system of 0 (absent disease) to 28 (severe disease) (high score indicative of poor quality of life [QOL]). Values after first rescue treatment used were set to missing (censoring) before MI.
Time Frame: Baseline through Week 36
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 83 | 84 | 86 | 169
units on a scale | 7.0 (0.90) | 2.8 (0.78) | 0.8 (0.73) | -0.3 (0.56)

14. Secondary Outcome: Absolute Change From Baseline in Dermatology Life Quality Index (DLQI) Through Week 36
Description: The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life (QOL). The 10 questions assessed QOL over the past week, with an overall scoring of 0 (absent disease) to 30 (severe disease); a high score was indicative of a poor QOL. Values after first rescue treatment used were set to missing before MI.
Time Frame: Baseline through Week 36
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 83 | 84 | 86 | 169
units on a scale | 3.1 (0.52) | 1.5 (0.46) | 0.3 (0.48) | -0.2 (0.33)

15. Secondary Outcome: Absolute Change From Baseline in Hospital Anxiety Depression Scale (HADS) Through Week 36
Description: HADS is a fourteen item scale. Seven of the items relate to anxiety and seven items relate to depression. Each item on the questionnaire is scored from 0 (minimum score) - 3 (maximum score) and this means that a person can score between 0 (no symptoms) and 21 (severe symptoms) for either anxiety or depression. Cut-offs for identifying psychiatric distress has been reported as 7 to 8 for possible presence, 10 to 11 for probable presence, and 14 to 15 for severe anxiety or depression. Values after first rescue treatment used were set to missing before MI.
Time Frame: Baseline through Week 36
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 83 | 84 | 86 | 169
units on a scale | 0.8 (0.60) | 0.7 (0.52) | 0.2 (0.54) | -0.8 (0.39)

16. Secondary Outcome: Difference Between Current Study Baseline and Week 36 in Percent Change in SCORAD From Parent Study Baseline
Description: SCORAD is a clinical tool for assessing the severity of AD developed by the European Task Force on Atopic Dermatitis (Severity scoring of atopic dermatitis: the SCORAD index). Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology (Basel) 186 (1): 23-31. 1993. Extent and intensity of eczema as well as subjective signs (insomnia, etc.) are assessed and scored. Total score ranges from 0 (absent disease) to 103 (severe disease). Values after first rescue treatment used were set to missing before MI.
Time Frame: Baseline (Parent Study), Baseline (Current Study) and Week 36 (Current study)
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 83 | 84 | 86 | 169
Percent change | 28.97 (3.683) | 10.42 (2.988) | 2.21 (2.743) | 0.33 (2.092)

17. Secondary Outcome: Difference Between Current Study Baseline and Week 35 in Percent Change in Peak Weekly Pruritus NRS From Parent Study Baseline
Description: as for outcome 11
Time Frame: Baseline (Parent Study), Baseline (Current Study) and Week 35 (Current study)
Population: FAS population was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 83 | 84 | 86 | 169
percent change | 35.6 (4.32) | 16.7 (4.09) | 8.6 (4.02) | -0.1 (3.05)

18. Secondary Outcome: Annualized Event Rate of Skin Infection Treatment- Emergent Adverse Events (TEAEs)
Description: Any untoward medical occurrence in a participant who received investigational medicinal product (IMP) was considered an AE without regard to possibility of causal relationship with this treatment. Treatment- emergent adverse events (TEAEs) were defined as AEs that developed or worsened or became serious during on- treatment period (time from the first dose of study drug up to the end of study [Week 36]). A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in any of the following outcomes: death, life- threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. Any TEAE included participants with both serious and non-serious AEs.
Time Frame: Baseline through Week 36
Population: FAS population was used.
Measure: Median (95% Confidence Interval); unit: events per year
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 83 | 84 | 86 | 169
events per year | 0.12 [0.044 to 0.338] | 0.07 [0.024 to 0.226] | 0.02 [0.005 to 0.120] | 0.02 [0.007 to 0.083]

19. Secondary Outcome: Annualized Event Rate of Flares
Description: Rate of Flares defined as worsening of disease requiring initiation or escalation of rescue treatment.
Time Frame: Baseline through week 36
Population: FAS population was used.
Measure: Median (95% Confidence Interval); unit: events per year
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 83 | 84 | 86 | 169
events per year | 0.75 [0.465 to 1.214] | 0.60 [0.363 to 0.977] | 0.39 [0.231 to 0.661] | 0.24 [0.146 to 0.380]

20. Secondary Outcome: Percentage of Well-Controlled Weeks During the On-treatment Period
Description: Well-controlled weeks are those in which participants during their weekly IVRS call completion has their eczema been well-controlled over the last week during which no rescue treatments were administered. Percentage of well-controlled weeks during the on-treatment period were reported.
Time Frame: Baseline through Week 36
Population: The safety analysis set (SAF) included all randomized participants who received any amount of study drug. Here, number of participants analyzed = participants with available data for this endpoint. One participant was randomized to Dupilumab Q2W/QW, but treated per Dupilumab Q4W arm and included in SAF.
Measure: Mean (Standard Deviation); unit: percentage of weeks
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
Number analyzed (Participants) | 81 | 82 | 87 | 165
percentage of weeks | 40.9 (30.35) | 53.2 (32.95) | 52.3 (35.96) | 63.6 (32.08)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (Week 36) regardless of seriousness or relationship to investigational product.
Description: Reported AEs are treatment-emergent adverse events that developed/worsened during the 'on-treatment period' (time from the first dose of study drug up to the end of study [Week 36]). The safety analysis set (SAF) included all randomized participants who received any amount of study drug. Note: One participant was randomized to Dupilumab Q2W/QW, but treated per Dupilumab Q4W arm and included in the SAF
Arm/Group | Placebo QW | Dupilumab 300 mg Q8W | Dupilumab 300 mg Q4W | Dupilumab 300 mg Q2W/QW
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/84 | 1/87 | 0/167
Serious Adverse Events (participants affected / at risk) | 1/82 | 3/84 | 4/87 | 6/167
Other Adverse Events (participants affected / at risk) | 55/82 | 43/84 | 47/87 | 72/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo QW (N=82) | Dupilumab 300 mg Q8W (N=84) | Dupilumab 300 mg Q4W (N=87) | Dupilumab 300 mg Q2W/QW (N=167)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia induced cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Open fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biochemical pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament Rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo QW (N=82) | Dupilumab 300 mg Q8W (N=84) | Dupilumab 300 mg Q4W (N=87) | Dupilumab 300 mg Q2W/QW (N=167)
Injection site reaction (General disorders) | 2 (22) | 3 (10) | 2 (8) | 10 (62)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 5 (6) | 3 (4)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 5 (7) | 4 (4)
Nasopharyngitis (Infections and infestations) | 11 (13) | 11 (14) | 11 (14) | 32 (41)
Oral herpes (Infections and infestations) | 3 (4) | 5 (10) | 2 (5) | 3 (10)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 7 (7) | 5 (6) | 13 (16)
Headache (Nervous system disorders) | 2 (6) | 3 (3) | 5 (7) | 8 (12)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 40 (60) | 27 (34) | 30 (43) | 34 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.